CLINICAL TRIAL: NCT00081055
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of OTI-010 in Subjects Who Receive HLA-Identical Sibling Peripheral Blood Stem Cell Transplantation for Hematologic Malignancies
Brief Title: OTI-010 for Graft-Versus-Host Disease Prophylaxis in Treating Patients Who Are Undergoing Donor Peripheral Stem Cell Transplantation for Hematologic Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast International Sàrl (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: Mesoblast; UCLA-0303036; CDR0000358809 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes
Keywords: graft versus host disease; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; refractory anemia; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Congenital Abnormalities | interventions — Busulfan; Cyclophosphamide; Cyclosporine; Methotrexate; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: autologous expanded mesenchymal stem cells OTI-010
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: OTI-010 may be effective for graft-versus-host disease prophylaxis (prevention) in patients who are undergoing donor peripheral stem cell transplantation for hematologic malignancies (cancer of the blood or bone marrow).

PURPOSE: This randomized phase II trial is studying how well OTI-010 works in preventing graft-versus-host disease in patients who are undergoing donor peripheral stem cell transplantation for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the safety and efficacy of OTI-010 vs placebo as graft-versus-host disease prophylaxis in patients with hematologic malignancies undergoing HLA-identical sibling matched peripheral blood stem cell transplantation.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to age (18 to 34 vs 35 to 55) and donor/recipient gender (female donor/male recipient vs female donor/female recipient vs male donor/female recipient vs male donor/male recipient).

* Conditioning regimen: Patients receive cyclophosphamide IV once daily on days -5 and -4 and undergo total body irradiation twice daily on days -3 to -1 OR busulfan IV over 2 hours every 6 hours on days -7 to -4 and cyclophosphamide IV once daily on days -3 and -2.
* Graft-versus-host disease prophylaxis: Patients receive methotrexate IV on days 1, 3, 6, and 11. Patients also receive cyclosporine orally or IV (over 1-4 hours) twice daily beginning on day -1 and continuing for at least 6 months followed by a taper until 1 year after transplantation.
* OTI-010 therapy: Patients are randomized to 1 of 3 treatment arms.

  * Arm I: Patients receive placebo IV 4 hours before peripheral blood stem cell transplantation (PBSCT) on day 0.
  * Arm II: Patients receive OTI-010 IV 4 hours before PBSCT on day 0.
  * Arm III: Patients receive a higher dose of OTI-010 IV 4 hours before PBSCT on day 0.
* Allogeneic stem cell transplantation: Patients undergo allogeneic PBSCT on day 0.

Patients are followed at 18 weeks, at 6, 9, and 12 months, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 99 patients (33 per treatment arm) will be accrued for this study within 5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following hematologic malignancies:

  * Acute lymphoblastic leukemia, meeting 1 of the following criteria:

    * In first or second remission
    * In early first or second relapse*
  * Acute myeloid leukemia, meeting 1 of the following criteria:

    * In first or second remission
    * In early first or second relapse*
  * Chronic myelogenous leukemia

    * Chronic or accelerated phase
  * Any of the following myelodysplastic syndromes:

    * Refractory anemia (RA)
    * RA with ringed sideroblasts
    * RA with excess blasts NOTE: *< 24% marrow blasts and < 5% peripheral blood blasts (within 10 days of beginning conditioning regimen)
* No secondary acute leukemia
* Prior CNS tumor involvement allowed provided patient is asymptomatic and there is no evidence of CNS disease on lumbar puncture and CT scan of the brain
* Must have a 6/6 HLA-identical sibling donor available

PATIENT CHARACTERISTICS:

Age

* 18 to 55

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)
* SGOT < 10 times ULN
* Hepatitis B core antigen, surface antigen, and e-antigen negative
* Hepatitis B DNA negative
* Hepatitis C RNA negative

Renal

* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* LVEF ≥ 50% by MUGA or echocardiogram
* No right sided heart failure

Pulmonary

* FEV_1 > 50% of predicted
* DLCO ≥ 50% of predicted (corrected for anemia)
* Oxygen saturation ≥ 97% on room air
* No pulmonary hypertension

Immunologic

* HIV-1 and 2 antibody negative
* HIV-1 antigen negative
* HTLV-I and II antibody negative
* No active infection

Other

* CNS function normal
* No uncontrolled alcohol or substance abuse within the past 6 months
* No other concurrent underlying medical condition that would preclude study participation
* Not pregnant
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior allogeneic or autologous hematopoietic stem cell transplantation
* No concurrent medication to accelerate neutrophil or platelet engraftment except filgrastim (G-CSF)

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No prior solid organ transplantation

Other

* More than 30 days since prior investigational agents or devices
* No other concurrent investigational agents or devices
* No concurrent anti-infective therapy except prophylactic therapy
* No other concurrent conditioning regimen agents
* No concurrent herbal remedies except multivitamins
* No other concurrent graft-versus-host disease prophylaxis medications (e.g., ursodeoxycholic acid)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Incidence of acute GVHD grade II-IV of skin, liver and gut (stomach to rectum) through Day 84 post-PBSC transplantation | Day 84

SECONDARY OUTCOMES:
Safety as measured by infusional toxicity, relapse nd survival, formation of potential ectopic tissue foci | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Mary C. Territo, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States